## Comparison of hydro-dissection versus ultrasonic aspirator in division of liver parenchyma in laparoscopic resection

**Lap Liver Study** 

NCT03208192

20/02/2017

## **CONSENT TO PARTICIPATE**

In prospective randomized single-center study: "Comparison of hydro-dissection versus ultrasonic aspirator in division of liver parenchyma in laparoscopic resection"

Principal Investigators: [Names]

Please initial the following as appropriate:

I have read and understood the information sheet on the above study and have had the opportunity to discuss the details with the researchers and ask questions. I had enough time to make this decision. At the moment I have no issues.

I have agreed to take part in the study as it has been outlined to me, but I understand that I am free to withdraw from the study or any part of the study at any time, without having to give a reason. My withdrawal will not lead to any unwanted consequences for my further treatment.

I understand that authorized representatives of regulatory agencies, and the Ethic Committee can see some sections of my medical records related to my participation in this study.

In case of withdrawal from the study or termination of a sponsor or researcher, I give my consent to the processing of my data collected to that time.

Transmission and storage of information is carried out in accordance with the Laws of the Russian Federation on the protection of confidential information.

In case of refusal from the further participation in the study, I agree that my data will be stored and analysed in accordance with the foregoing, in the case of availability, can be used in similar studies.

I hereby fully and freely give my informed consent to take part in this study.

| lame of participant: |
|---------------------------|
| Signature of participant: |
| )ate: |